CLINICAL TRIAL: NCT04417270
Title: Reliability of the Freestyle Libre CGM in the Inpatient Setting During the COVID-19 Surge
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwell Health (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 20-0455
Record Dates: First submitted 2020-06-01; First posted 2020-06-04 (Actual); Last update posted 2021-03-02 (Actual); Status verified 2021-03

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: Patients will use the Freestyle 14 day CGM reader or their phone to check their glucose. A clinical staff member will check the patient's blood sugar by performing a glucose finger stick with the Accuchek inform II meter.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Freestyle Libre 14-day CGM (Other): The FreeStyle Libre 14 day system is a continuous glucose monitoring system consisting of a handheld reader and a sensor worn on the back of the upper arm.
  Interventions: Device: Freestyle Libre 14 day CGM system; Device: Accuchek Inform II platform
- Accuchek Inform II meter (Other): ACCU-CHEK INFORM II system quantitatively measures glucose in fresh venous, arterial, neonatal heel stick and capillary whole blood from the finger and is used as an aid in monitoring the effectiveness of glucose control
  Interventions: Device: Freestyle Libre 14 day CGM system; Device: Accuchek Inform II platform

INTERVENTIONS:
Device: Freestyle Libre 14 day CGM system — The FreeStyle Libre 14 day system is a continuous glucose monitoring system consisting of a handheld reader and a sensor worn on the back of the upper arm.
Device: Accuchek Inform II platform — The Accu-Chek Inform II system is designed to deliver data with speed and efficiency, helping to provide optimal care. Wireless meter quickly transfers data. The Accu-Chek Inform II system is the first point-of-care blood glucose device to offer truly wireless technology at the meter level.

SUMMARY:
The FDA has provided an emergency waiver for the use of non-invasive continuous glucose monitors (CGM) in hospitals, so frontline health care providers (in hospitals) can remotely monitor patients with diabetes thus reducing patient's discomfort, limiting exposure to COVID-19 and preserving critical personal protective equipment (PPE). The FreeStyle Libre 14-day system is a continuous glucose monitoring system consisting of a handheld reader (smart phone may be used) and a sensor applied with adhesive to back of the upper arm. In order to evaluate the reliability of the Freestyle Libre CGM for in-patient use, we propose a study which will examine the correlation between the libre CGM data and capillary blood glucose test - the current standard of care taken by the Accuchek Inform II platform.

DETAILED DESCRIPTION:
In hospitalized patients diagnosed with COVID-19, diabetes mellitus is associated with a higher mortality. Patients with controlled blood glucose have a lower mortality rate than those who are uncontrolled. However, a rigid blood glucose control - which may lead to hypoglycemia- is associated with higher mortality rates. Thus, adequate glucose monitoring is important for hospitalized diabetic patients.

Previous studies have shown that CGMS, in the outpatient setting, engender better glycemic control thereby reducing risk of hypoglycemia. CGMS offer a replacement for finger stick blood glucose monitoring which may not identify an incidence of hypoglycemia until symptoms drive the patient to test. Furthermore, finger stick blood glucose monitoring is painful and time consuming thus causing many patients to avoid this aspect of diabetes self-care management.

Freestyle Libre CGMs sample interstitial fluid glucose subcutaneously. Measurement frequencies typically range from 1 to 15 minutes and most commonly are every 5 minutes.

Previous studies in hospitalized patients living with diabetes mellitus on basal bolus regimen have shown:

• Use of the CGM increased detection of both hypoglycemic and hyperglycemic events versus those sensed by POCT.

One investigation identified 88 postprandial hyperglycemic excursions in patients with CGM use as opposed to 61 in those with POCT. Another noted that when comparing the CGM use with that of POCT, the former identified 55 hypoglycemic events whereas the latter only found 12.

• No difference in mean daily glucose CGM and POCT readings. In a study of 38 patients, the investigators noted no difference in mean daily glucose between the CGM and POCT.

ELIGIBILITY:
Inclusion Criteria:

* Participants acquired from among all non-critical care in patients who are living with Diabetes Mellitus. Because the patients will have to be instructed on the use of the CGM, this study will be limited to English speaking/reading adults (18 years of age or older), who possess the cognitive and physical ability to participate.

Exclusion Criteria:

* Minors, pregnant women, and critically ill.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2020-06-12 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Comparison of values between two devices | Through end of patient hospitalization, an average of 14 days
  Correlation between blood glucose results from the Freestlye Libre 14-day CGM and Accuchek Inform II platform using the Bland-Altman method to determine whether the two glucose methods agree

CONTACTS AND LOCATIONS:
Overall Officials: Renee Murray-Bachmann, Ed.D, MSN, Principal Investigator — Northwell Health
Locations (1):
- Lenox Hill Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
The team has not decided whether to share the results with other researchers. The team will consider publishing results after study completion

REFERENCES:
- See also: Flash Glucose-Sensing Technology as a Replacement for Blood Glucose Monitoring for the Management of Insulin-Treated Type 2 Diabetes: A Multicenter, Open-Label Randomize — http://doi.org/10.1007/s13300-016-0223-6
- See also: Zhu, L., Zhi-Gang, S., Cheng, S., Guo, J., Bing-Hong, Z.,Hongliang, L. (2020).Association of blood glucose control and outcomes in patients with COVID-19 and pre-existing Type 2 Diabetes Cell Metabolism, 31, (2020).pp.1-10 — http://doi.org/10.1016/j.cmet.2020.04.021
- See also: Continuous Glucose Monitoring in the Hospital Panel (2017). Consensus Statement on Inpatient Use of Continuous Glucose Monitori — http://doi.org/10.1177/1932296817706151